CLINICAL TRIAL: NCT04421885
Title: An Open-Label, Randomized, Single-Dose, Semi-Replicate, 4-Period, Crossover, Bioequivalence Study Comparing Two Tablet Formulations of Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) in Healthy Adult Subjects
Brief Title: Bioequivalence Study Comparing Two Tablet Formulations of Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SPR994-105
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Open-Label, Randomized, Single-Dose, Semi-Replicate, 4-Period, Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A: TBPM-PI-HBr (Reference - fasted) (Experimental): 600 mg (2 x 300 mg tablets) clinical study drug product batch TBPM-PI-HBr administered at Hour 0 on Day 1, under fasted conditions.
  Interventions: Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) - Reference
- B: TBPM-PI-HBr (Test - fasted) (Experimental): 600 mg (2 x 300 mg tablets) registration drug product batch TBPM-PI-HBr administered at Hour 0 on Day 1, under fasted conditions.
  Interventions: Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) - Test
- C: TBPM-PI-HBr (Test - fed) (Experimental): 600 mg (2 x 300 mg tablets) registration drug product batch TBPM-PI-HBr administered at Hour 0 on Day 1, under fed conditions.
  Interventions: Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) - Test

INTERVENTIONS:
Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) - Reference — 600 mg (2 x 300 mg tablets) clinical study drug product batch TBPM-PI-HBr.
  Arms: A: TBPM-PI-HBr (Reference - fasted)
Drug: Tebipenem pivoxil hydrobromide (TBPM-PI-HBr) - Test — 600 mg (2 x 300 mg tablets) registration drug product batch TBPM-PI-HBr.
  Arms: B: TBPM-PI-HBr (Test - fasted); C: TBPM-PI-HBr (Test - fed)

SUMMARY:
A bioequivalence and food-effect study comparing two tablet formulations of tebipenem pivoxil hydrobromide (TBPM-PI-HBr) in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, 18 to 55 years of age
* Continuous non-smoker.
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs.
* Has suitable venous access for repeated blood sampling.
* A female of childbearing potential must agree to abstain from sexual activity that could lead to pregnancy.
* A female of non-childbearing potential.
* Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected to have during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease.
* History of any illness that might confound the results of the study or poses an additional risk to the subject by their participation in the study.
* History of significant allergic disease requiring treatment.
* History or presence of alcoholism or drug abuse.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
* History of known genetic metabolism anomaly associated with carnitine deficiency.
* Female subjects with a positive pregnancy test or who are lactating.
* Positive urine drug or alcohol results.
* Positive results for human immunodeficiency virus (HIV 1 and 2), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
* QTcF interval is > 460 msec (males) or > 470 msec (females) or has ECG findings deemed abnormal with clinical significance by the PI or designee at the screening visit.
* Estimated creatinine clearance < 80 mL/min at the screening visit.
* Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Area under the curve extrapolated to infinity (AUC0-∞). | 24h (Day 2) post dose (Arms: A, B, C)
Area under the concentration-time curve, from time 0 to the last observed non-zero concentration (t) (AUC0-t). | 24h (Day 2) post dose (Arms: A, B, C)
Maximum plasma concentration (Cmax). | 24h (Day 2) post dose (Arms: A, B, C)

SECONDARY OUTCOMES:
Time to the maximum plasma concentration (Tmax). | 24h (Day 2) post dose (Arms: A, B, C)
Terminal elimination half-life (t½). | 24h (Day 2) post dose (Arms: A, B, C)
Apparent total body clearance (CL/F) | 24h (Day 2) post dose (Arms: A, B, C)
Apparent volume of distribution during the terminal elimination phase after oral (extravascular) administration (Vz/F). | 24h (Day 2) post dose (Arms: A, B, C)
Incidence of treatment-emergent AEs (including SAEs) categorized by severity and relationship to study drug. | 12 to 14 days after the last dose of study drug
  ECG, Clinical Laboratories, Vitals Signs and Physical Exams will be used as a safety measure to detect any AEs.
Area under the curve extrapolated to infinity (AUC0-∞). | 24h (Day 2) post dose (Arms: B, C)
  TPBM PK parameters following administration of the TBPM-PI-HBr Test tablet under fasted and fed conditions.
Area under the concentration-time curve, from time 0 to the last observed non-zero concentration (t) (AUC0-t). | 24h (Day 2) post dose (Arms: B, C)
  TPBM PK parameters following administration of the TBPM-PI-HBr Test tablet under fasted and fed conditions.
Maximum plasma concentration (Cmax). | 24h (Day 2) post dose (Arms: B, C)
  TPBM PK parameters following administration of the TBPM-PI-HBr Test tablet under fasted and fed conditions.
Time to the maximum plasma concentration (Tmax). | 24h (Day 2) post dose (Arms: B, C)
  TPBM PK parameters following administration of the TBPM-PI-HBr Test tablet under fasted and fed conditions.
Terminal elimination half-life (t½). | 24h (Day 2) post dose (Arms: B, C)
  TPBM PK parameters following administration of the TBPM-PI-HBr Test tablet under fasted and fed conditions.
Apparent total body clearance (CL/F) | 24h (Day 2) post dose (Arms: B, C)
  TPBM PK parameters following administration of the TBPM-PI-HBr Test tablet under fasted and fed conditions.
Apparent volume of distribution during the terminal elimination phase after oral (extravascular) administration (Vz/F). | 24h (Day 2) post dose (Arms: B, C)
  TPBM PK parameters following administration of the TBPM-PI-HBr Test tablet under fasted and fed conditions.

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, Study Director — Spero Therapeutics
Locations (1):
- Medical Facility, Tempe, Arizona, United States